CLINICAL TRIAL: NCT06458049
Title: Sexual Health and Rehabilitation Online (SHAREonline): An Educational Intervention for Young Adult Women After Cancer
Brief Title: Sexual Health and Rehabilitation Online (SHAREonline)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sharon Bober, Ph.D, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-697; R21CA279278 (NIH)
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cancer Survivorship; Sexual Function Disturbances
Keywords: Cancer Survivorship; Sexual Function Disturbances
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHAREonline (Experimental): Participants will receive:
  * One online group session structured around three 60-minute modules and creation of a personal action plan
  * Single Coaching phone call at one month
  * Questionnaires to complete at baseline, 2 and 4 Months
  Interventions: Behavioral: Group Session; Behavioral: Coaching Call
- Individual Self Management (Active Comparator): Brief individualized session with online and written materials and guidance.
  All Participants will complete study questionnaires at baseline, 2 months and 4 months post intervention
  Interventions: Behavioral: Educational Materials

INTERVENTIONS:
Behavioral: Group Session — On-line educational session-3 modules-1 hour each for a total of 3 hours
  Arms: SHAREonline
Behavioral: Coaching Call — Single Coaching phone call at one month
  Arms: SHAREonline
Behavioral: Educational Materials — Individual videoconference session in which participants will receive a pdf of the American Cancer Society booklet, 'Sex and the Adult Female with Cancer
  Arms: Individual Self Management

SUMMARY:
SHAREonline is a study for young female cancer survivors that are experiencing changes in sexual health and function.

The purpose of this research is to compare two brief interventions delivered by videoconference to learn if they help women effectively manage these changes and restore sexual health and functioning.

DETAILED DESCRIPTION:
The purpose of this research is to compare two brief interventions delivered by videoconference to learn if they help women effectively manage these changes and restore sexual health and functioning.

Participants in this study would first complete health questionnaires and then be randomized to take part in one of two types of education sessions delivered by an instructor over videoconference: 1) Group education session or 2) Individual self-management session.

About 56 women will receive the group education session and about 28 will receive the individual self-management session.

It is expected that about 84 women will take part in this study.

ELIGIBILITY:
* Female cancer survivors age 19-49
* Cancer diagnosis (except non-melanoma skin cancer) ≥ 1 year prior
* Diagnosed with first cancer ≥ age 18
* No active cancer therapy (excluding chemoprevention) in the past four months, and no further therapy planned
* Ability to read and write in English
* Bothered by significant sexual dysfunction as evidenced by a Female Sexual Functioning Index (FSFI) score of ≤26.
* Regular access to the internet

Exclusion Criteria

* Has never been sexually active
* Any impairment (e.g., hearing, visual, cognitive) that interferes with the ability to complete all study procedures independently

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual Function | Baseline to 2 months
  The Female Sexual Function Index (FSFI Full Scale Score), is 19-item instrument which measures sexual function, including desire, orgasm, pain and satisfaction.

SECONDARY OUTCOMES:
Change in Emotional Distress | Baseline to 2 month
  BSI-18 (Brief Symptom Inventory) The BSI-18 is a well-validated screening measure of psychological distress with subscales measuring anxiety, depression and somatization that is frequently used with oncology populations.
Change in Sexual Function | Baseline to 4 months
  The Female Sexual Function Index (FSFI Full Scale Score), is 19-item instrument which measures sexual function, including desire, orgasm, pain and satisfaction.
Change in Emotional Distress | Baseline to 4 months
  BSI-18 (Brief Symptom Inventory) The BSI-18 is a well-validated screening measure of psychological distress with subscales measuring anxiety, depression and somatization that is frequently used with oncology populations.
Enrollment Rate | Baseline to 1 month
  Measured through study accrual with a benchmark of enrollment greater than or equal to 40% of eligible candidates
Intervention Acceptability Rate | Up to 1 month-post intervention
  Intervention Satisfaction Questionnaire will be assessed using a benchmark mean score of 4
Study Engagement Rate | Baseline to 1 month
  Measured through study engagement with a benchmark of study engagement greater than or equal to 70% of eligible candidates
Intervention Completion Rate | Baseline to 4 months
  Measured through intervention completion with a benchmark of intervention completion greater than or equal to 60% of eligible candidates
Distress about Sexual Function | Baseline to 2 months
  Sexual Distress Scale-short form (SDS-SF) is a 5-item measure which assesses distress about sexual function.
Distress about Sexual Function | Baseline to 4 months
  Sexual Distress Scale-short form (SDS-SF) is a 5-item measure which assesses distress about sexual function.
Sexual Function, Satisfaction and Sexual Inactivity | Baseline to 2 months
  PROMIS Sexual Function and Satisfaction (PROMIS SexFS) is a short screening

OTHER OUTCOMES:
Sexual Self-efficacy | Baseline to 2 months
  Sexual Self-Efficacy Scale is a 5-item scale developed to measure perceived sexual self-efficacy to address sexual health after cancer.
Sexual Self-efficacy | Baseline to 4 months
  Sexual Self-Efficacy Scale is a 5-item scale developed to measure perceived sexual self-efficacy to address sexual health after cancer.
Coaching Satisfaction Summary | Up to 1 month post-coaching session
  Brief participant questionnaire to provide feedback about coaching session.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Bober, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu